CLINICAL TRIAL: NCT01140074
Title: Effectiveness and Efficacy of Zinc With Probiotics for the Treatment of Acute Diarrhea in Young Children
Brief Title: Efficacy of Zinc Sulfate With Probiotics for the Treatment of Acute Diarrhea in Children
Acronym: Zinc
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital No 1 Wroclaw (Other)
Responsible Party: prof Leszek Szenborn, Katedra i Klinka Pediatrii i Chorob Infekcyjnych AM we Wroclawiu
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: KB-501/2009
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Acute Watery Diarrhoea
Keywords: acute diarrhoea, children
MeSH Terms: interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc sulfate (Experimental): Children in active treatment group will be given zinc sulfate 10-20 mg per day orally plus probiotics
  Interventions: Drug: Zinc Sulfate
- Placebo (Placebo Comparator): Children will be given placebo plus probiotics
  Interventions: Drug: Zinc Sulfate

INTERVENTIONS:
Drug: Zinc Sulfate — Zinc Sulfate in sugar sirup will be given orally in dosis of 10-20 mg per day for 10 days
  Other Names: brand product is not available in Poland

SUMMARY:
Diarrheal disease is one of the major causes of morbidity and mortality in children under five. Disease is treated symptomatically with oral rehydration (ORS) as a basic measure. In children with severe zinc deficiency, diarrhea is common and responds quickly to zinc supplementation. Zinc supplementation may also helpful in diarrheal children without zinc deficiency. Effectiveness of zinc was proven in developing countries but was not in Europe. Objective of our study is to assess whether zinc supplementation given with probiotics and ORS is effective in acute diarrhea in children in Poland.

DETAILED DESCRIPTION:
A double-blind, placebo controlled trial

- We are going to enroll 256 patients (aged > 1 months to 36 months) with acute watery diarrhea defined as 3 d or more watery stools per day lasting not less than 1 day and not longer than 5 days.

Exclusion criteria:

severe dehydration (> 10%) Coexisting severe infection (E.g. Sepsis, pneumonia, meningitis) Immune deficiency Chronic digestive tract disease (e.g. celiac diseases, food allergy) Therapy with Antibiotics

Patients will be randomly assigned to 2 groups to receive: (a) zinc sulfate 10-20 mg/day for 10 days plus probiotics for 5 days (b) placebo for 10 days plus probiotics for 5 days. Patients will be observed in ambulatory or in the hospital (if necessary) and followed up for 15 days.

Randomization 1:1

ELIGIBILITY:
Inclusion Criteria:

* Age 1-36 months
* Acute diarrhea defined as 3 or more watery stools per day
* Informed consent (parents)

Exclusion Criteria:

* Severe dehydration (> 10%)
* Coexisting severe infection (e.g. sepsis, pneumonia, meningitis)
* Immune deficiency
* Chronic digestive tract disease (e.g. celiac diseases, food allergy)
* Antibiotic therapy

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Period of diarrhea in hours | 15 days
  The primary endpoint of our study is the time of acute diarrhea

SECONDARY OUTCOMES:
number of stools in consequent days | 15 days
  The secondary end points will be number of stools per day, necessity of hospitalization or not, tolerability and adherence to the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Szenborn, Prof, Principal Investigator — Wroclaw Medical University
Locations (2):
- Poland (2):
  - Szpital im Sw Jadwigi w Trzebicy, Trzebnica
  - Klinika Pediatrii i Chorob Infekcyjnych Akademii Medycznej we Wroclawiu, Wroclaw

REFERENCES:
- [Background] Larson CP, Nasrin D, Saha A, Chowdhury MI, Qadri F. The added benefit of zinc supplementation after zinc treatment of acute childhood diarrhoea: a randomized, double-blind field trial. Trop Med Int Health. 2010 Jun;15(6):754-61. doi: 10.1111/j.1365-3156.2010.02525.x. Epub 2010 Mar 29. PMID 20374562
- [Background] Fajolu IB, Emokpae A, Oduwole AO, Silva BO, Abidoye RO, Renner JK. Zinc supplementation in children with acute diarrhoea. Nig Q J Hosp Med. 2008 Apr-Jun;18(2):101-3. doi: 10.4314/nqjhm.v18i2.44997. PMID 19068562
- [Background] Boran P, Tokuc G, Vagas E, Oktem S, Gokduman MK. Impact of zinc supplementation in children with acute diarrhoea in Turkey. Arch Dis Child. 2006 Apr;91(4):296-9. doi: 10.1136/adc.2005.079939. Epub 2005 Dec 14. PMID 16354711
- [Result] Roy SK, Tomkins AM, Akramuzzaman SM, Behrens RH, Haider R, Mahalanabis D, Fuchs G. Randomised controlled trial of zinc supplementation in malnourished Bangladeshi children with acute diarrhoea. Arch Dis Child. 1997 Sep;77(3):196-200. doi: 10.1136/adc.77.3.196. PMID 9370894